CLINICAL TRIAL: NCT05574933
Title: Racism-based Stress Injury and Biomarkers of Stress: A Feasibility Study and Correlation Study
Brief Title: Racism-based and Biomarkers of Stress
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: RKI-1036
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Racism; Stress, Psychological
MeSH Terms: conditions — Racism; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for a complete blood count, gene expression analysis, and telomere length testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This feasibility study aims to explore how racism-induced stress impacts the brain and body and how a culturally responsive intervention can reduce the mental and physical effects of this stress among African Americans (AA). We aim to acquire methodological and protocol insights for a subsequent study by assessing 1) the feasibility of recruiting AA for a race-related study and collecting psychological and biomarkers of stress, 2) determining the association between racism-based stress surveys and biomarkers of stress, and 3) explore participants feedback on the impact of racism in their life and their willingness to participate in a 12-week mindfulness intervention with additional assessments, such as functional MRI testing.

DETAILED DESCRIPTION:
Racism is a chronic stressor affecting minority groups, particularly Black, Indigenous, and People of Color (BIPOC), which increases their vulnerability to disease and adverse outcomes. Several studies have associated racism with psychosocial distress, elevated inflammation, and accumulation of toxic radicals in the body, leading to diabetes and heart disease. Moreover, studies investigating biological structural changes suggest that racism is associated with alterations in activation and connectivity of brain regions controlling emotional behavior. Race-based encounters can lead to high levels of stress that can cause a traumatic reaction raising chronic vigilance by creating anticipatory distress and concerns, which could drive the output of allostatic mediators. Allostatic load represents the cumulative physiological burden exacted on the body throughout a lifetime in the effort to adapt to stressors. Therefore, in addition to broader structural and institutional changes, there is a critical need for interventions to mitigate race-related injury and promote enhanced physical and mental health.

Contemplative-Based Resilience Training (CBRT) is a potential non-invasive intervention that may moderate the effects of racism on health outcomes. CBRT is a contemplative self-healing program that integrates mindfulness with cognitive education, affect modulation, motivational imagery, breath control, and self-massage. Research demonstrates that compassion-based meditative therapies support the development of pro-social attributes and social connections. Individuals with higher mindfulness traits are thought to have a greater ability to regulate their emotions and are less emotionally reactive. In addition, mindfulness interventions can also lead to the development of individual resilience and by focusing on the present moment, negative feelings are less likely to persist leading to psychological well-being and consequently physiological health. Mindfulness-based interventions are efficacious in reducing anxiety, depression, substance abuse, eating disorders, and chronic pain and improving general well-being and quality of life. Although there is some evidence of the buffering effect of mindfulness on psychological outcomes from discrimination, few studies have focused on race-based stress and are limited to examining psychological outcomes.

This feasibility study aims to acquire methodological and protocol insights and build the infrastructure for a subsequent CBRT interventional study to reduce the effects of race-based trauma and stress. The study will be a mixed-methods study with an embedded qualitative study. First, we will determine if it is feasible to recruit a sample of 20 African American/Black participants to measure behavioral and physiological measures of race-based stress. Second, we will validate and further test additional physiological variables of racism as a stressor on allostatic load, gene expression, and telomere length. Third, we will conduct interviews to obtain participants' perspectives and feedback on a planned 12-week mindfulness intervention study to reduce the effects of race-based stress among African Americans, as well as to assess their willingness to undergo additional assessments, such as functional MRI scans. The deliverables of this study are to build a community-based research infrastructure, to determine with greater clarity some of the relationships between physiological variables and racism-induced stress, and how to adapt an existing CBRT intervention to address the experience of race-based stress in a more culturally responsive manner.

ELIGIBILITY:
Inclusion Criteria:

* Self Identity as African American or Black
* 18-50 years old
* Fluent in English
* Born and or raised in the United States

Exclusion Criteria:

* History of significant pre-existing brain disease or injury (e.g., dementia, stroke, seizure disorder, and head injury with cognitive sequelae or loss of consciousness >30 min.ute, seizure disorder)
* Reported history of learning disability/mental retardation
* Current Attention Deficit Hyperactive Disorder (ADHD), depression, bipolar disorder, post-traumatic stress disorder (PTSD), or psychotic disorder diagnosis
* Current psychotropic medication (as these medications have known impacts on brain function) eg. antipsychotics, antianxiety
* Severe/chronic medical illness (e.g., reported HIV+ status, cardiovascular disease, liver disease/cirrhosis, chronic kidney disease, current/past cancer with radiation/chemotherapy treatment, etc.)
* Current methadone/suboxone/buprenorphine (or similar) maintenance
* Use of illicit substances other than cannabis within the past 90 days
* Pregnant
* Major life events in the last 30 days (hospitalization, marriage, death in the family of friends, disaster)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Self-identifying African Americans/Black 18-50 years of age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of study | 2 weeks
  percentage of participants who complete the study
Correlation analysis of race-based traumatic stress and allostatic load | 2 weeks
  Correlate levels of race-based traumatic stress calculated from a questionnaire (Race-based Traumatic stress symptoms-RBTSSS) with allostatic load and stress biomarkers (salivary cortisol). The RBTSS is 52 items self-report instrument that assesses reactions resulting from negative racial experiences. Participants identify the most memorable negative racial encounter and complete emotional symptom reaction items. Items are rated along a 5-point Likert scale. RBTSSS comprises of 7 symptom scales: Depression (10 items), Intrusion (8 items), Anger (8 items), hypervigilance (8 items), physical reactions (8 items), Low self-esteem (6 items), and avoidance (4 items). Higher scores indicate a greater presence of reaction symptoms. The Allostatic score is calculated as a composite of 10 biomarkers focused on the metabolic, renal, and immune physiologic systems.
Acceptability of planned 12 week intervention | 2 weeks
  Percentage of participants willing to participate in a future planned Intervention

SECONDARY OUTCOMES:
Allostatic load composite score | 2 weeks
  The Allostatic score was calculated as a composite of these 10 biomarkers focused on the metabolic, renal, and immune physiologic systems. A Biomarkers from the metabolic system included body mass index (BMI) (kg/m2), albumin, and alkaline phosphatase. The renal system biomarkers were creatinine and creatinine clearance, and immune system biomarkers were C-reactive protein (CRP) and white blood cell count (WBC). The cut points are determined by pre-established values in clinical medicine and generate three categories: high-risk (1 point), moderate-risk (0.5 point), and low-risk (0 points)
Telomere Length | 2 weeks
  Quantitative RT-PCR will be used to determine average telomere length
Salivary Cortisol-AUC | After baseline, 3 timepoints at waking, 30min after waking, and at bedtime. In a 24 hour period
  Samples will be collected using the passive drool technique using a . Participants will be instructed to gather saliva samples 3 times in one day: at waking, 30min after waking, and at bedtime. Participants will be instructed not to eat, drink or brush their teeth during the 30 min prior to sample collection times. Salivary cortisol will be analyzed using area-under-the-curve (AUC)
Concentrations of pro-inflammatory gene expression Response to Adversity (CTRA) | 2 weeks
  Gene expression measures of immune system function will be collected via Paxegene tubes. Analyses will focus on a priori-specified gene regulation pattern involving increased expression of inflammation-related genes and decreased expression of antiviral genes - a pattern called the conserved transcriptional response to adversity
Qualitative evaluation of participants perspectives on racism based stress | 2 weeks
  Qualitative interviews using semistructured questions will be conducted to understand participants' perspectives on racism and how they cope with racism
Race-based traumatic stress symptoms | 2 weeks
  Race-based Traumatic stress symptoms (RBTSSS) is a 52-item self-report instrument that assesses reactions resulting from negative racial experiences. Participants identify the most memorable negative racial encounter and complete emotional symptom reaction items. Items are rated along a 5-point Likert scale. RBTSSS comprises of 7 symptom scales: Depression (10 items), Intrusion (8 items), Anger (8 items), hypervigilance (8 items), physical reactions (8 items), Low self-esteem (6 items), and avoidance (4 items). Higher scores indicate a greater presence of reaction symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel W Kimani, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Public Health Association. Analysis: Declarations of Racism as a Public Health Crisis.2021. https://www.apha.org/-/media/Files/PDF/topics/racism/Racism_Declarations_Analysis. ashx
- [Background] Williams DR, Mohammed SA. Racism and Health I: Pathways and Scientific Evidence. Am Behav Sci. 2013 Aug 1;57(8):10.1177/0002764213487340. doi: 10.1177/0002764213487340. PMID 24347666
- [Background] Bailey ZD, Krieger N, Agenor M, Graves J, Linos N, Bassett MT. Structural racism and health inequities in the USA: evidence and interventions. Lancet. 2017 Apr 8;389(10077):1453-1463. doi: 10.1016/S0140-6736(17)30569-X. PMID 28402827
- [Background] Becares L, Nazroo J, Kelly Y. A longitudinal examination of maternal, family, and area-level experiences of racism on children's socioemotional development: Patterns and possible explanations. Soc Sci Med. 2015 Oct;142:128-35. doi: 10.1016/j.socscimed.2015.08.025. Epub 2015 Aug 15. PMID 26301485
- [Background] Paradies Y, Ben J, Denson N, Elias A, Priest N, Pieterse A, Gupta A, Kelaher M, Gee G. Racism as a Determinant of Health: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 23;10(9):e0138511. doi: 10.1371/journal.pone.0138511. eCollection 2015. PMID 26398658
- [Background] Geronimus AT, Hicken M, Keene D, Bound J. "Weathering" and age patterns of allostatic load scores among blacks and whites in the United States. Am J Public Health. 2006 May;96(5):826-33. doi: 10.2105/AJPH.2004.060749. Epub 2005 Dec 27. PMID 16380565
- [Background] Clark US, Miller ER, Hegde RR. Experiences of Discrimination Are Associated With Greater Resting Amygdala Activity and Functional Connectivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Apr;3(4):367-378. doi: 10.1016/j.bpsc.2017.11.011. Epub 2017 Dec 8. PMID 29628069
- [Background] Akdeniz C, Tost H, Streit F, Haddad L, Wust S, Schafer A, Schneider M, Rietschel M, Kirsch P, Meyer-Lindenberg A. Neuroimaging evidence for a role of neural social stress processing in ethnic minority-associated environmental risk. JAMA Psychiatry. 2014 Jun;71(6):672-80. doi: 10.1001/jamapsychiatry.2014.35. PMID 24740491
- [Background] Brody GH, Lei MK, Chae DH, Yu T, Kogan SM, Beach SRH. Perceived discrimination among African American adolescents and allostatic load: a longitudinal analysis with buffering effects. Child Dev. 2014 May-Jun;85(3):989-1002. doi: 10.1111/cdev.12213. Epub 2014 Feb 5. PMID 24673162
- [Background] Epel ES, Blackburn EH, Lin J, Dhabhar FS, Adler NE, Morrow JD, Cawthon RM. Accelerated telomere shortening in response to life stress. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17312-5. doi: 10.1073/pnas.0407162101. Epub 2004 Dec 1. PMID 15574496
- [Background] Thomas MD, Sohail S, Mendez RM, Marquez-Magana L, Allen AM. Racial Discrimination and Telomere Length in Midlife African American Women: Interactions of Educational Attainment and Employment Status. Ann Behav Med. 2021 Jun 28;55(7):601-611. doi: 10.1093/abm/kaaa104. PMID 33289498
- [Background] Tull ES, Sheu YT, Butler C, Cornelious K. Relationships between perceived stress, coping behavior and cortisol secretion in women with high and low levels of internalized racism. J Natl Med Assoc. 2005 Feb;97(2):206-12. PMID 15712783
- [Background] Miller HN, LaFave S, Marineau L, Stephens J, Thorpe RJ Jr. The impact of discrimination on allostatic load in adults: An integrative review of literature. J Psychosom Res. 2021 Jul;146:110434. doi: 10.1016/j.jpsychores.2021.110434. Epub 2021 Mar 24. PMID 33810863
- [Background] Watson-Singleton NN, Pennefather J, Trusty T. Can a culturally-responsive Mobile health (mHealth) application reduce African Americans' stress?: A pilot feasibility study. Current Psychology. 2021 /03/02 2021;doi:10.1007/s12144-021-01534-9
- [Background] Carter RT, Muchow C. Construct validity of the Race-Based Traumatic Stress Symptom Scale and tests of measurement equivalence. Psychol Trauma. 2017 Nov;9(6):688-695. doi: 10.1037/tra0000256. Epub 2017 Feb 6. PMID 28165267
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Wei M, Alvarez AN, Ku TY, Russell DW, Bonett DG. Development and validation of a Coping with Discrimination Scale: factor structure, reliability, and validity. J Couns Psychol. 2010 Jul;57(3):328-44. doi: 10.1037/a0019969. PMID 21133583
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649